CLINICAL TRIAL: NCT00913575
Title: Effect of Pre-surgery Neuromuscular Physiotherapy (PT) on Functional Outcome After Total Knee Replacement (TKR): A Single-blinded Randomized Controlled Trial.
Brief Title: Effect of Pre-surgery Neuromuscular Physiotherapy (PT)
Acronym: Omega
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Olten (Other); Kantonsspital Aarau (Other); Lund University (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Erika Huber, ex. MHSA, PT, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/012
Record Dates: First submitted 2009-05-12; First posted 2009-06-04 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Knee Osteoarthritis
Keywords: neuromuscular training; preoperative exercise; physiotherapy; total knee replacement; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preoperative neuromuscular training (Experimental): preoperative neuromuscular training
  Interventions: Other: preoperative neuromuscular training
- education (Placebo Comparator): knee school
  Interventions: Behavioral: knee OA School

INTERVENTIONS:
Other: preoperative neuromuscular training — The neuromuscular training group will receive a minimum of 8 and a maximum of 24 training sessions; as well as 4 sessions of the Knee OA School.
  Other Names: exercise
  Arms: preoperative neuromuscular training
Behavioral: knee OA School — The education group will only receive 4 sessions of the Knee OA School.
  Other Names: knee school
  Arms: education

SUMMARY:
Background:

Osteoarthritis (OA) is a common degenerative condition of large weight-bearing joints, such as the hip and knee, as well as small hand joints. Current interventions in patients with OA are limited to symptomatic pain relief and later with total joint replacement (TJR). While TJR improves function and pain, it does not fully restore function in most individuals. A key factor of functional outcome is probably conditioning before and after TJR surgery. However, this has not been studied conclusively in patients undergoing TKR surgery.

Objective:

1. Primary endpoint: To study the effect of a pre-surgery neuromuscular PT compared to an attention control program on lower extremity function measured by the Chair stands test (observed function) and the KOOS score (reported function).
2. Secondary endpoints will be muscle strength, walking time and mobility.

Hypothesis:

The investigators hypothesize that patients undergoing pre-surgery PT will be significantly quicker in performing the chair stands test and report a significant improvement in the KOOS at 3 months after surgery compared to controls.

Methods:

80 patients from a waiting list for unilateral TKR will be randomized to neuromuscular PT or an attention control group intervention in a single-blinded randomized controlled trial. Assessments will be at baseline, at 3 months after surgery and at 12 months after surgery.

Intervention:

The neuromuscular PT group will receive a minimum of 8 and a maximum of 24 training sessions; all patients, including the control group, will receive 4 sessions of the Knee School.

Significance:

Given the demographic change with an increase in the older segment of the population there will be a rise in the absolute number of TKRs. It is therefore warranted to study pre-surgery neuromuscular PT to help patients get the most out of their joint replacement.

DETAILED DESCRIPTION:
Due to the demographic change with a significant increase in the older segment of the population, recent estimates in the United States suggest that the rate of TKR surgery will rise exponentially over the next decade. A similar trend is expected in Switzerland with a marked increase in the absolute number of TKR surgery. Today, patients waiting for TKR surgery in Switzerland are neither routinely participating in an active training program to reduce pain and improve function nor in an educational program to increase coping skills before surgery.

The intervention group will receive neuromuscular training as well as 4 sessions of the Knee OA School. Both will be offered in group sessions separate from the control group.

a) The neuromuscular training will take place under the supervision of an experienced physiotherapist, 2 sessions a week of 60 minutes each. The training program, based on neuromuscular and biomechanical principles, according to the possibilities of the patient. The training sessions consists of three parts: warming up (ergometer cycling), a circuit program, and cooling down (walking, stretching, mobility). The circuit program comprises four exercise circles with the key elements of core stability, postural function, functional alignment, lower extremity muscle strength, and functional exercises.

b) The Knee School is an educational program and takes place in three group sessions and one individual follow-up session. Patients receive information about: anatomy and physiology of the knee (first group session); proposed physical activity and pain self-management (second group session); and the rehabilitation phase after surgery (third group session).

The control group will receive the Knee School sessions without the neuromuscular PT separate from the intervention group to avoid interaction between the groups.

ELIGIBILITY:
Inclusion criteria:

* Primary TKR for primary or secondary OA
* Age 60 years or older
* Community-dwelling
* German language skills in word and writing

Exclusion criteria:

* Age older than 85 years
* Cognitive impairment
* Revision surgery
* Plan to leave Switzerland before or/and after surgery
* History of inflammatory arthritis
* Unable to walk for at least 3 meters with or without walking aid

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Lower limb function by the Chair stands (observed measure) | 6 wks pre-surgery, 1 wk pre-surgery 3 months post-surgery

SECONDARY OUTCOMES:
Lower limb function by the Knee Injury and Osteoarthritis Outcome Score (KOOS) (observed measure) | 6 wks pre-surgery, 1 wk pre-surgery, 6 wks post-surgery, 3 months post-surgery, 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heike A Bischoff-Ferrari, MD, DrPH, Principal Investigator — UniversitaetsSpital Zuerich, Switzerland; Ewa M Roos, PT, Prof Dr, Principal Investigator — University of Southern Denmark, Denmark; Rob A de Bie, PT, Prof Dr, Principal Investigator — Maastricht University, Netherlands; Christoph A Schwaller, MD, Dr, Principal Investigator — Kantonsspital Olten; Marc Zumstein, MD, Dr, Principal Investigator — Kantonsspital Aarau, Switzerland
Locations (1):
- University Hospital, Centre on Aging and Mobility, Zurich, Switzerland

REFERENCES:
- [Derived] Huber EO, de Bie RA, Roos EM, Bischoff-Ferrari HA. Effect of pre-operative neuromuscular training on functional outcome after total knee replacement: a randomized-controlled trial. BMC Musculoskelet Disord. 2013 May 3;14:157. doi: 10.1186/1471-2474-14-157. PMID 23641782